CLINICAL TRIAL: NCT00671814
Title: A Double-Blind, Placebo and Active Controlled, Single and Multiple Rising Dose, Safety, Tolerance, and Pharmacokinetic Study of TR-701 in Normal Healthy Adults
Brief Title: Single and Multiple Ascending Dose Pharmacokinetic Study of TR701 in Healthy Adults
Acronym: SAD/MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1986-016; TR701-101 (Other: TriusRX Unique ID)
Record Dates: First submitted 2008-05-01; First posted 2008-05-05 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Healthy Subjects
Keywords: antibiotic
MeSH Terms: interventions — tedizolid phosphate; Linezolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Single oral dose of TR-701 given once at 200mg, 400mg, 600mg, 800mg, and 1200mg. Multiple oral doses of TR-701 given once daily for 21 days at 200mg, 300mg and 400mg.
  Interventions: Drug: TR-701
- 2 (Placebo Comparator): Single oral dose of placebo given in cohorts 1-5. Multiple oral doses of placebo given once daily for 21 days in cohorts 6-8 and twice daily for 21 days in cohort 10.
  Interventions: Drug: placebo
- 3 (Active Comparator): Oral doses of 600mg linezolid given twice daily for 21 days.
  Interventions: Drug: linezolid

INTERVENTIONS:
Drug: TR-701 — TR-701 will be given as single oral doses in Cohorts 1-5 and as once daily oral doses for 21 days in cohorts 6-8.
  Arms: 1
Drug: linezolid — Linezolid will be given at 600 mg twice daily for 21 days in cohort 10.
  Arms: 3
Drug: placebo — Placebo will be given once for cohorts 1-5, once daily for 21 days for cohorts 6-8, and twice daily for 21 days for cohort 10.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of single rising oral doses and multiple oral doses of TR-701

DETAILED DESCRIPTION:
This is an evaluation of TR-701 in a double-blind, placebo-controlled, randomized, single (Part A) and multiple (Part B) ascending dose safety, tolerance, and PK when administered as a capsule in normal, healthy adult volunteers. The study will be sequential between Part A and Part B (i.e., not staggered or leap frogged), with slight overlap between last cohort in Part A and first cohort in Part B.

ELIGIBILITY:
Inclusion Criteria:

* in good health
* body mass index of 20 to 29.9 kg/m2
* female subjects must be either postmenopausal for at least 1 year, surgically sterile, abstinent, or agree to use an effective method of birth control

Exclusion Criteria:

* history or clinical manifestations of any clinically significant disorder
* history of hypersensitivity or allergies to any drug compound
* history of stomach or intestinal surgery or resection
* history of alcoholism or drug addiction within 1 year
* use of any tobacco-containing or nicotine-containing products within 6 months
* use of any other medications
* use of alcohol-containing, grapefruit-containing, or caffeine-containing foods or beverages; or foods or beverages with high levels of tyramine
* pregnancy, lactation, or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-01-06 (Actual); Primary Completion 2008-06-06 (Actual); Study Completion 2008-06-06 (Actual)

PRIMARY OUTCOMES:
Adverse Event reporting | 21 days

SECONDARY OUTCOMES:
The PK rate and extent of urinary excretion of TR-701 and its microbiologically active moiety, TR-700 | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: John Bohn, MD, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Lodise TP, Bidell MR, Flanagan SD, Zasowski EJ, Minassian SL, Prokocimer P. Characterization of the haematological profile of 21 days of tedizolid in healthy subjects. J Antimicrob Chemother. 2016 Sep;71(9):2553-8. doi: 10.1093/jac/dkw206. Epub 2016 Jun 17. PMID 27317442
- [Derived] Flanagan SD, Bien PA, Munoz KA, Minassian SL, Prokocimer PG. Pharmacokinetics of tedizolid following oral administration: single and multiple dose, effect of food, and comparison of two solid forms of the prodrug. Pharmacotherapy. 2014 Mar;34(3):240-50. doi: 10.1002/phar.1337. Epub 2013 Aug 7. PMID 23926058